CLINICAL TRIAL: NCT00518856
Title: Lufwanyama Neonatal Survival Project
Acronym: LUNESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Tufts University (Other)
Responsible Party: Davidson H. Hamer, Boston University School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GHS-A-00-03-00020-00-4
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Mortality
Keywords: birth asphyxia; neonatal sepsis; maternal to child transmission of HIV
MeSH Terms: conditions — Asphyxia Neonatorum; Neonatal Sepsis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): TBAs who receive training and supplies for the intervention
  Interventions: Other: Neonatal resuscitation protocol
- control (Active Comparator): TBAs continuing with current standard of practice
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Neonatal resuscitation protocol — training in neonatal resuscitation and sepsis identification early treatment
  Arms: intervention
Other: Standard of care — continued with current standard of care for birth attendants
  Arms: control

SUMMARY:
We seek to determine whether we can reduce day 28 mortality in Zambian newborns by training traditional birth attendants a modified version of the neonatal resuscitation protocol (NRP) and by improving their abiltiy to identify sepsis and initiate antibiotics in the field.

DETAILED DESCRIPTION:
This is a cluster randomized trial of the impact of providing additional training and supplies to traditional birth attendants in a rural setting in Zambia. 120 TBAs are randomized into intervention/control. Intervention TBAs receive NRP training, supplies for neonatal resuscitation, receiving blankets for thermoregulation, and amoxicillin tablets. Control TBAs continue according to prior standard of care. Primary outcome is mortality at 28 days life as a proportion of births attended by TBAs in each study arm.

ELIGIBILITY:
Inclusion Criteria:

* TBA trained in safe delivery;
* willing to sign informed consent; willing to be randomized; willing to adhere to study procedures

Exclusion Criteria:

* TBA living outside of Lufwanyama district

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3559 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
mortality | day 28

SECONDARY OUTCOMES:
perinatal mortality | day zero
sepsis mortality | deaths between days 1-28
cost effectiveness | days 0-28
successful delivery of nevirapine prophylaxis to HIV exposed deliveries | day zero umbilical cord dried blood spot

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Gill, MD MS, Principal Investigator — Boston Universtiy; Grace Mazala, RN, Study Director — Lufwanyama District Health Management Team

REFERENCES:
- [Derived] Gill CJ, Guerina NG, Mulenga C, Knapp AB, Mazala G, Hamer DH. Training Zambian traditional birth attendants to reduce neonatal mortality in the Lufwanyama Neonatal Survival Project (LUNESP). Int J Gynaecol Obstet. 2012 Jul;118(1):77-82. doi: 10.1016/j.ijgo.2012.02.012. Epub 2012 Apr 27. PMID 22542215
- [Derived] Gill CJ, Phiri-Mazala G, Guerina NG, Kasimba J, Mulenga C, MacLeod WB, Waitolo N, Knapp AB, Mirochnick M, Mazimba A, Fox MP, Sabin L, Seidenberg P, Simon JL, Hamer DH. Effect of training traditional birth attendants on neonatal mortality (Lufwanyama Neonatal Survival Project): randomised controlled study. BMJ. 2011 Feb 3;342:d346. doi: 10.1136/bmj.d346. PMID 21292711